CLINICAL TRIAL: NCT00005812
Title: A Pilot Phase II Trial of Temozolomide in Leptomeningeal Metastases
Brief Title: Temozolomide in Treating Patients With Leptomeningeal Metastases From a Solid Tumor or Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No objective response documented, protocol terminated after 12 patients.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9812; DMS-9812; NCI-G00-1782
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Brain Tumors; Central Nervous System Tumors; Leptomeningeal Metastases
Keywords: leptomeningeal metastases; temozolomide
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Meningeal Carcinomatosis | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental): Oral temozolomide 75 mg/m2/day for 6 weeks, followed by 4 week break. Cycles will continue until:
  * disease progression
  * intolerable toxicity
  * complete response - 2 full additional cycles
  * if response is complete except for residual radiographic abnormalities that persist unchanged for 2 full cycles: continue for 4 cycles past best response.
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients who have leptomeningeal metastases from a solid tumor or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate, survival time, and quality of life of patients with leptomeningeal metastases from a solid tumor or lymphoma when treated with oral temozolomide.
* Determine adverse events related to this regimen in this patient population.
* Measure temozolomide concentrations in CSF and serum and correlate with appropriate pharmacodynamic parameters (e.g., response) in these patients.

OUTLINE: Patients receive oral temozolomide daily for 6 weeks. Courses repeat every 10 weeks in the absence of unacceptable toxicity or disease progression.

Patients with a complete response (CR) receive 2 additional courses after achieving CR. Patients with a CR except for residual radiographic abnormalities that persist unchanged for 2 full courses continue for 4 courses past best response.

Quality of life is assessed at baseline, weekly for the first 4 weeks of therapy, and then monthly thereafter.

PROJECTED ACCRUAL: A total of 14-24 patients will be accrued for this study.

ELIGIBILITY:
* Documented leptomeningeal metastases
* Carcinomatous meningitis that is previously untreated or failed prior therapy OR
* Lymphomatous meningitis
* Systemic disease that is responding or stable on current therapy not eligible if discontinuing therapy would be deleterious
* Age 18 and over
* Karnofsky Performance Status 60-100%
* Life expectancy of at least 6 weeks
* Absolute neutrophil count greater than 1,500/μL
* Platelet count greater than 100,000/μL
* Creatinine no greater than 2.0 mg/dL
* No congestive heart failure
* No unstable angina
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindication to diagnostic sampling of CSF via lumbar puncture or reservoir
* No medical conditions that would interfere with absorption of oral medication (e.g., malabsorption, obstruction, or frequent vomiting)
* No uncontrolled infection
* Prior neuroaxis chemotherapy (lumbar puncture, reservoir, or systemic) allowed
* No other concurrent chemotherapy for other sites of disease
* No prior radiotherapy to areas of measurable meningeal disease unless there is clear radiographic progression in these areas
* No prior radiotherapy to greater than 30% of bone marrow
* Prior radiotherapy to the neuroaxis allowed
* No concurrent radiotherapy for other sites of disease or for progressive disease
* Recovered from any prior recent therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-01; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Objective Response | Every 6 weeks
  Response will be assessed clinically, cytologically, and radiographically.

SECONDARY OUTCOMES:
Pharmacokinetics | Every 6 weeks
  Drug levels in cerebrospinal fluid assessed every 6 weeks
Survival | every 6 weeks
Quality of Life | Baseline, weekly during cycle 1, before each additional cycle
  FACT-Br

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H. Davis, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Davis TH, Fadul CE, Glantz MJ, et al.: Pilot phase II trial of temozolomide for leptomeningeal metastases: preliminary report. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-460, 2003. ISBN 1932312021